CLINICAL TRIAL: NCT05300776
Title: A Multi-center Prospective Clinical Study of M-ROSE Combined With mNGS to Guide the Individualized Anti-infection Treatment, Prevention and Control of Drug-resistant Bacteria in Severe Hospital-acquired Pneumonia
Brief Title: M-ROSE Combined With mNGS in Severe Hospital-acquired Pneumonia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Beijing Anzhen Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, wang kaifei, Clinical Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: shoufa2022-1-5091
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Pneumonia
Keywords: M-ROSE; mNGS; severe hospital-acquired pneumonia; treatment
MeSH Terms: conditions — Pneumonia; Healthcare-Associated Pneumonia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-ROSE combined with mNGS group (Experimental): The bronchoalveolar lavage fluid (BALF) of patients undergoes M-ROSE analysis and decide whether the samples are qualified, whether they indicate bacterial infection and identify pathogens, and the qualified samples are sent for mNGS analysis. The individualized anti-infection treatment is comprehensively guided according to the results of M-ROSE, mNGS and clinical examinations.
  Interventions: Diagnostic Test: M-ROSE analysis
- mNGS group (No Intervention): BALF samples were directly sent for mNGS analysis, and anti-infective treatment was guided according to clinical examinations.

INTERVENTIONS:
Diagnostic Test: M-ROSE analysis — The M-ROSE analysis process consists of 3 procudures.
  1. Specimen quality assessment. The BALF undergoes the process of smear, diff-quik stain, gram stain and are analyzed by experts to report the cytoloy and pathogen patterns to determine whether the sample is qualified according to the cell proportions. The qualified BALF samples are: squamous epithelial cell proportion<1%, columnar epithelial cell proportion <5% .
  2. Distinguish infection and colonization. According to the cytoloy pattern, the proportion of neutrophils > 50% often strongly suggests pulmonary bacterial infection; Neutrophil phagocytosis proportion> 5% indicates infection, and phagocytosis of bacteria is the pathogen. Besides, fungal and hyphae can be found under the microscope.
  3. Preliminary identification of infectious pathogens. Identify the infected bacteria and fungi, and the results are gram-positive cocci, gram-positive bacilli, gram-negative cocci, gram-negative bacilli, yeasts and molds.
  Arms: M-ROSE combined with mNGS group

SUMMARY:
The purpose of this study is to determine the value of M-ROSE（microbiological rapid on-site evaluation）in severe hospital-acquired pneumonia.

DETAILED DESCRIPTION:
Severe hospital acquired pneumonia (SHAP) is the critical risk factor leading to the death of nosocomial infection patients. Rapid identification of pathogens, guidance of individualized treatment and rational application of antibiotics can not only improve the administration of antibiotics, but also reduce the production of multi drug resistant bacteria. Metagenomic second-generation sequencing (mNGS) is an important tool to quickly identify the pathogen in ICU. However, due to the low qualified rate of lower respiratory tract specimens in patients with SHAP, easily polluted, and the difficulty to determine whether microorganisms are infectious, colonizated or polluted, the value of mNGS was limited in the etiological diagnosis of SHAP. The bedside M-ROSE system established by our research team can determine whether the lower respiratory tract specimen is qualified, whether infection exists and the pathogen of infection within half an hour. Based on the previous work, this project plans to conduct a prospective multicenter, single blind, randomized controlled study under the guidance of M-ROSE and mNGS in the individualized anti-infection strategy of SHAP, to reduce the mortality of patients with SHAP; Combined with the third-generation sequencing, the standard analysis framework for the traceability and prevention and control of drug-resistant bacteria was established to clarify the transmission route of drug-resistant bacteria, so as to provide a new solution for the prevention and control of clinical multidrug-resistant bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe hospital-acquired pneumonia
* Must have undergone bronchoalveolar lavage

Exclusion Criteria:

* BALF samples were not sent for mNGS examination
* Age < 18 years old
* The hospitalization days ≤ 3
* The clinical data are incomplete
* Mechanical ventilation time > 60 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
mortality | During the intervention.
  Alive or Dead.

SECONDARY OUTCOMES:
Blood leukocyte ratio tread | During the intervention.
  The changing of blood leukocyte ratio
28 day outcome | 28 days after admission
  Live or dead.
Blood neutriphil ratio tread | During the intervention.
  The changing of blood neutriphil ratio tread
Blood interleukin 6 tread | During the intervention.
  The changing of blood interleukin 6 tread
Blood C-reactive protein | During the intervention.
  The changing of blood C-reactive protein
Blood procalcitonin tread | During the intervention.
  The changing of blood procalcitonin tread

CONTACTS AND LOCATIONS:
Overall Officials: Lixin Xie, Ph.D, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Yi Tao, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Wang K, Xie F, Han Z, Liu Y, Pan L, Zhu G, Cao Z, Yan P, Xiao L, Duan Z, Hu Y, Xiao K, Chen X, Fu H, Shi Y, Song Y, Han X, Xie W, Xie L. Protocol of a multicenter, single-blind, randomized, parallel controlled trial evaluating the effect of microbiological rapid on-site evaluation (M-ROSE) guiding anti-infection treatment in patients with severe hospital-acquired pneumonia. Trials. 2023 Aug 23;24(1):552. doi: 10.1186/s13063-023-07570-z. PMID 37612723